CLINICAL TRIAL: NCT06540898
Title: The Effects of Mindful Eating and Movement on Food Literacy, Physical Literacy and Social Emotional Competencies Among University Students in Macau
Brief Title: Impact of Mindful Eating and Movement on University Students' Food and Physical Literacy, and Social-Emotional Competencies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Macau (Other)
Responsible Party: Principal Investigator, Siman Lei, Assistant Professor, University of Macau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE-0138-2024
Record Dates: First submitted 2024-07-24; First posted 2024-08-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Mindful Eating; Mindful Movement; Food Literacy; Physical Literacy; Social-Emotional Learning; Health Behavior; Nutrition
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Participants in this arm engage in an 8-week program that integrates mindful eating and mindful movement practices into their regular physical education classes. Each class includes a 10-minute mindful eating practice focused on enhancing awareness of hunger and fullness cues, sensory experiences of food, and emotional responses to eating. Following this, the final 10 minutes of each class are dedicated to mindful movement exercises, which combine physical postures and movement with mindfulness techniques to promote food literacy, physical literacy and social emotional competencies.
  Interventions: Behavioral: Mindfulness-Based Eating and Movement Program
- Control Group (No Intervention): Standard Physical Education Participants in this arm continue with their regular physical education classes as usual, without the integration of any mindfulness practices. This control arm involves the standard activities and curriculum designed for physical education classes at the university, which may include a variety of physical exercises, sports, and theoretical instruction related to health and fitness.

INTERVENTIONS:
Behavioral: Mindfulness-Based Eating and Movement Program — This intervention integrates mindful eating practices and mindful movement into physical education classes for a duration of 8 weeks.
  Each session begins with a 10-minute mindful eating practice designed to enhance participants; awareness of hunger and fullness cues, the sensory experience of eating, and their emotional responses to food. The program is to address food literacy, physical literacy, and social-emotional learning. It applied the principles of various established mindfulness and cognitive behavioral therapies and the book "The Joy of Half a Cookie: Using Mindfulness to Lose Weight and End the Struggle with Food" . It is grounded in the components of Mindfulness-Based Eating Awareness Training. The movement practices include basic poses in pairs and groups, and breath awareness techniques to facilitate a mindful connection with physical sensations and mental states.
  Arms: Experimental Group

SUMMARY:
The goal of this clinical trial is to investigate if the mindful eating and movement program can improve food literacy, physical literacy, and social-emotional competencies in university students aged 18-25 years. The main questions it aims to answer are:

1. Will the mindful eating and movement program lead to significant improvements in food literacy?
2. Will the mindful eating and movement program enhance physical literacy?
3. Will the mindful eating and movement program improve social-emotional competencies?

Researchers will compare an intervention group receiving the combined mindful practices with a control group participating in standard physical education to see if the intervention group shows greater improvements in these areas.

Participants will:

Engage in mindful eating exercises during the break of physical education classes for 10 minutes.

Participate in mindful movement exercises before each physical education class end for 10 minutes, in pairs or in groups.

Complete baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after) assessments to measure changes in food literacy, physical literacy, and social-emotional competencies.

ELIGIBILITY:
Inclusion Criteria:

1. University undergraduate students aged 18 to 25 years old who are not pregnant;
2. Chinese-speaking adults;
3. Willing to sign the consent form;
4. Willing to attend mindful practice regularly;
5. No prior experience with formal mindfulness practices such as mindful eating or mindful movement.

Exclusion Criteria:

1. Not university undergraduate students;
2. Below 18 years old or above 25;
3. Non-Chinese speaking adults;
4. Unable or refuse to sign the consent form;
5. Refuse to attend mindful practice regularly;
6. History of eating disorders;
7. Severe mental health disorders requiring ongoing treatment;
8. Physical conditions limiting participation in physical activities.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Food Literacy Evaluation Questionnaire (FLEQ-Ch) | Baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after).
  Improvement in food literacy knowledge will be assessed using the Food Literacy Evaluation Questionnaire (FLEQ-Ch). This 15-item questionnaire is structured into three main dimensions: Planning and Management, Selection, and Preparation. It evaluates participants' knowledge related to making informed food choices. Participants respond to each item using a 4-point Likert scale ranging from 0 (Never) to 3 (Always). The total score ranges from 0 to 45, with higher scores indicating higher levels of food literacy.
Mindful Eating Questionnaire (MEQ) | Baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after).
  Improvement in mindful eating behaviors will be assessed using the Mindful Eating Questionnaire (MEQ), designed by Framson et al. (2009). This 28-item questionnaire evaluates eating behavior across five subscales: Awareness, Distraction, Disinhibition, Emotional Response, and External Cues. Participants rate a 4-point Likert scale from 1 (never/rarely) to 4 (usually/always). The total MEQ score is calculated as the average of all subscale scores, ranging from 28 to 112. The higher the score, the higher degree of mindful eating behavior.
24-Hour Dietary Intake Records | Baseline, each mindfulness session, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after).
  Improvement in food literacy will be assessed through 24-hour dietary intake records. This metric evaluates participants' ability to maintain balanced eating habits. The 24-hour dietary intake will be measured each time on the day of the mindfulness session and on the days when participants complete the questionnaires.
Perceived Physical Literacy Instrument (PPLI) | Baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after).
  Enhancement in physical literacy will be assessed using the Perceived Physical Literacy Instrument (PPLI). This instrument consists of 9 items across three subscales: Knowledge and Understanding, Self-Expression and Communication with Others, and Sense of Self and Self-Confidence. The Knowledge and Understanding subscale evaluates participants' attitudes and awareness of the health benefits of sports. The Self-Expression and Communication with Others subscale evaluates participants' social skills and confidence in natural environments. The Sense of Self and Self-Confidence subscale evaluates participants' physical fitness and self-management skills. The instrument consists of 9 items that are rated on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). The total score for the PPLI ranges from 9 to 45, with higher scores indicating higher levels of perceived physical literacy.
International Physical Activity Questionnaire (IPAQ-SF) | Baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after).
  Enhancement in physical activity levels will be assessed using the International Physical Activity Questionnaire (IPAQ-SF). This metric evaluates the frequency and duration of various physical activities over the past 7 days. It contains of 7 items. The total score for the IPAQ-SF is calculated in Metabolic Equivalent of Task (MET) minutes per week, reflecting the energy expenditure for each type of activity. The minimum score is 0 MET-minutes per week, indicating no physical activity, while there is no fixed maximum score, as it depends on the reported duration and frequency of activities. Higher scores on the IPAQ-SF indicate higher levels of physical activity, reflecting greater energy expenditure.
International Fitness Scale (IFIS) | Baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after).
  Enhancement in self-reported fitness elements will be assessed using the International Fitness Scale (IFIS). This metric evaluates participants' general fitness, cardiorespiratory fitness, muscle strength, speed and agility, and flexibility (1 = very poor, 2 = poor, 3 = average, 4 = good, 5 = very good). IFIS consists of 5 items, the total score is the sum of the individual item scores ranging from 5 to 25. Higher scores represent better perceived physical fitness across the different dimensions assessed.
Social and Emotional Competencies Questionnaire (SEC-Q) | Baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after).
  Development in social-emotional competencies will be assessed using the Social and Emotional Competencies Questionnaire (SEC-Q), developed by Zych et al. (2018). This 16-item questionnaire measures social-emotional competencies across four dimensions: Self-awareness, Self-management and Motivation, Social Awareness and Prosocial Behavior, and Decision-making. Each item rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score is calculated by summing all subscale scores, from 16 to 80. The higher the score, the greater the social and emotional competence.
Social Emotional Learning Scale-Young Adult Form (SELS-YF) | Baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after).
  Measured using the Social Emotional Learning Scale-Young Adult Form (SELS-YF), developed by Karacan-Özdemir and Büyükçolpan (2021). This 20-item questionnaire measures the social-emotional learning skills of individuals aged 18-24 across five dimensions based on the Collaborative for Academic, Social, and Emotional Learning (CASEL) model (2003): Self-awareness, Academic self-regulation, Social awareness, Relationship-building skills, and Responsible decision-making skills. Participants rated on a 5-point Likert scale from 1 (never) to 5 (always). Total scores range from 20 to 100, The higher the score, the greater the social-emotional learning skills.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale Short Form (DERS-SF) | Baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after).
  Improvement in emotional regulation will be assessed using the Difficulties in Emotion Regulation Scale Short Form (DERS-SF). This metric evaluates participants' abilities to regulate their emotions effectively. Participants rate each item on a 5-point Likert scale, indicating how often the items apply to them, from 1 (almost never) to 5 (almost always). Each subscale score is computed as the sum of its corresponding items, with the total DERS-SF score calculated by summing all 18 items. This results in a range from 18 to 90, with higher scores indicating greater difficulties in emotion regulation.
Perceived Stress Scale (PSS-10) | Baseline, immediately post-intervention (8 weeks), and one month post-intervention (4 weeks after)
  Reduction in stress levels will be assessed using the Perceived Stress Scale (PSS-10). This metric evaluates the degree to which participants perceive their lives as unpredictable, uncontrollable, and overloaded. Each question scores from 0 (never) to 4 (very often). Questions 1 to 3 are assessed using a direct scoring method, whereas questions 4 to 8 are evaluated using a reverse scoring method. The total PSS-10 score is calculated by adding up the scores of each item, with individual scores ranging from 0 to 40. Greater scores correspond to greater levels of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: SiMan LEI, Doctoral, Principal Investigator — University of Macau
Locations (2):
- Macau (2):
  - UM Sports Complex (N8) , Avenida da Universidade Taipa, Macau, China, Macao
  - University of Macau, Macao

IPD SHARING:
Plan to Share IPD: No